CLINICAL TRIAL: NCT00871962
Title: Long-term Oxygen Treatment (LTOT) in Chronic Obstructive Pulmonary Disease: Factors Influencing Survival: Survival Factors in COPD Treated by Long-term Oxygen Therapy
Brief Title: Long-term Oxygen Treatment (LTOT) in Chronic Obstructive Pulmonary Disease: Factors Influencing Survival
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Association Nationale pour les Traitements A Domicile, les Innovations et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: ANTADIR 2009 - COHORTE
Record Dates: First submitted 2009-03-27; First posted 2009-03-30 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: long-term oxygen therapy; COPD patients on necessity of long-term oxygen therapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood gaz analysis
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: COPD patients on necessity of long-term oxygen therapy
  Interventions: Other: OXYGEN SUPPLEMENTATION

INTERVENTIONS:
Other: OXYGEN SUPPLEMENTATION — Patients treated by LTOT, with or without clinically fulfilled criteria for LTOT, with PaO2<55mmHg or less at rest or during sleeping or less during exercise, if supplemental oxygen is demonstrated to improve the exercise-associated hypoxia. Patients with PaO2 56-59mmHg if they also have dependent edema, pulmonary hypertension or hematocrit higher than 56%
  Other Names: Patients with LTOT: survival

SUMMARY:
The purpose of this prospective cohort study is to determine factors involved in survival in new COPD patients treated by long-term oxygen therapy.

Background: long-term oxygen therapy is indicated in patients with severe COPD. No studies have been performed in the past 20-25 years to examine the results of early clinical trials. Further studies are necessary to understand the utility of oxygen therapy in severe COPD.

DETAILED DESCRIPTION:
long-term oxygen therapy prolongs life in patients with severe COPD and severe resting hypoxemia. The objective of this study is to measure the survival in relation to the level of initial resting hypoxemia, serious co-morbidities, and nutritional status in COPD patients treated by long-term oxygen therapy. After enrollment at the beginning of oxygen therapy, following data will be collected during 3 years. Lung function, blood gas analysis, exercise capacity measured by the 6-Min Walk Distance test (6-MWD), dyspnea scale, BODE index, quality of life, indirect and direct costs will be analyzed every year.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients on necessity of long-term oxygen therapy
* Patients treated by LTOT, with or without clinically fulfilled criteria for LTOT, with PaO2<55mmHg or less at rest or during sleeping or less during exercise, if supplemental oxygen is demonstrated to improve the exercise-associated hypoxia. Patients with PaO2 56-59mmHg if they also have dependent edema, pulmonary hypertension or hematocrit higher than 56%
* Patient clinically stable
* Patient with oxygen device of ANTADIR network
* Oral and written consent

Exclusion Criteria:

* Patient with obstructive sleep apnea or overlap syndrome
* Patient with non invasive ventilation
* Patient with evolutive cancer.
* Inability to complete questionnaires
* Inability to attend outpatient clinic

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients on necessity of long-term oxygen therapy
Sampling Method: Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2009-06; Primary Completion 2015-12 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Survival in function of initial hypoxemia, body mass index and cardiovascular events | 3 years

SECONDARY OUTCOMES:
Long-term oxygen therapy observance and duration | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: MELLONI Boris, Pr, Principal Investigator — Association Nationale pour les Traitements A Domicile, les Innovations et la Recherche
Locations (1):
- Service de Pneumologie, Hôpital du Cluzeau, Limoges, France